CLINICAL TRIAL: NCT06461897
Title: A Phase 3, Open-label, Efficacy-Assessor-Blinded Study, Comparing the Safety and Efficacy of Upadacitinib to Dupilumab in Children From 2 to Less Than 12 Years of Age With Moderate to Severe Atopic Dermatitis
Brief Title: A Study to Assess Adverse Events and Change in Disease Activity Comparing Oral Upadacitinib to Subcutaneous Dupilumab in Children From 2 to Less Than 12 Years of Age With Moderate to Severe Atopic Dermatitis
Acronym: Start Up
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M17-380; 2023-504713-76-00 (Other: EU CT)
Record Dates: First submitted 2024-06-12; First posted 2024-06-17 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis; Upadacitinib; RINVOQ
MeSH Terms: conditions — Dermatitis, Atopic | interventions — upadacitinib; dupilumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dupi-IR Cohort (Experimental): Participants in this cohort will receive upadacitinib medium dose.
  Interventions: Drug: Upadacitinib
- Randomized Cohort (Experimental): Participants in the Randomized Cohort will be randomized to receive either medium dose upadacitinib daily adult equivalent dose, low dose upadacitinib daily adult equivalent dose or dupilumab every 2 weeks or 4 weeks (at the label-indicated dose and frequency).
  Interventions: Drug: Upadacitinib; Drug: Dupilumab

INTERVENTIONS:
Drug: Upadacitinib — Oral Tablet or Oral Solution
  Other Names: ABT-494; RINVOQ®; RINVOQ LQ
Drug: Dupilumab — Subcutaneous Injection
  Arms: Randomized Cohort

SUMMARY:
Atopic dermatitis (AD) is a skin condition that may cause a rash and itching due to inflammation of the skin. Topical therapies applied over the skin may not be enough to control the AD in trial participants who require systemic anti-inflammatory treatment. This study compares upadacitinib to dupilumab in pediatric participants with moderate to severe AD who are candidates for systemic therapy. Adverse events and change in the disease activity will be assessed.

Upadacitinib is an approved drug for treating AD patients aged 12 or older. Participants will receive upadacitinib (given as daily dose) or dupilumab (given at label indicated dose every 2 or 4 weeks). Participants will be stratified depending on disease severity, age and response to previous treatment. There is 1 in 5 chance for participants to receive dupilumab during the randomized cohort. Approximately 675 participants aged 2 to less than 12 years of age will be enrolled in this study at approximately 150 sites worldwide. The study population (As defined by participants age or prior treatment) to be enrolled in the study is dependent on local regulatory requirement and/or agreement.

Participants will receive upadacitinib oral tablets once daily (or oral solution twice a day) for 160 weeks, or dupilumab as per its label for 52 weeks, and followed for 30 days after the last dose of upadacitinib and at least 12 weeks after the last dose of dupilumab.

There may be higher treatment burden for participants in this trial compared to their standard of care . Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by clinical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* A minimum weight of 10 kg and weight and height > 5th percentile for their age according to local standard growth charts at the Baseline Visit.
* Atopic Dermatitis (AD), according to Hanifin and Rajka criteria, with onset of symptoms at least 6 months prior to Baseline.
* Eczema Area and Severity Index (EASI) score >= 16; vIGA-AD score >= 3 (Note: In countries where dupilumab is only approved for severe AD, subjects to be included in the Randomized Cohort should have severe AD [vIGA-AD = 4]); >= 10% Body Surface Area of AD involvement at the Baseline Visit; and Baseline weekly average of daily Worst Itch Scale (WIS) or Worst Scratch/Itch numerical rating scale (WSI-NRS) >= 4.
* Participant must satisfy at least one of the following criteria (Note: More than 1 criterion may apply to an individual participant. All applicable criteria for each individual participant should be reported):
* To be included in the Randomized Cohort (Note: Participants must have severe AD [vIGA-AD = 4] in countries where dupilumab is approved only for severe AD.):

  1. [For all countries except US] Documented history of inadequate response or intolerance to TCS and/or TCI OR for whom use of one or more of these topical treatments is medically inadvisable (e.g., high disease burden, Scoring Atopic Dermatitis (SCORAD) > 50, EASI score > 21, or vIGA-AD > 3).
  2. For dupilumab-naïve participants: History of inadequate response to a systemic therapy for AD other than dupilumab or oral corticosteroids or for whom the available systemic treatments are otherwise medically inadvisable (e.g., because of important side effects or safety risks).
  3. History of inadequate response to 2 or more courses of oral corticosteroid therapy given for >= 14 days within 6 months prior to Screening or history of oral corticosteroid rebound, defined as recurrence of AD symptoms within 4 months after its discontinuation.
  4. For dupilumab-exposed participants: Prior exposure to dupilumab without documented history of inadequate response or intolerance (i.e., discontinuation of dupilumab for a non-medical reason, such as, but not limited to, non-coverage or loss of coverage for the drug by health insurance, or other logistic challenges [not safety- or efficacy-related] precluding the participants continued access to dupilumab).
* To be included in the Dupi-IR/Dupi-Medically Inadvisable Cohort:

  * Previous inadequate response or intolerance to dupilumab OR
  * Dupilumab is medically inadvisable (e.g., allergy to a component of dupilumab, etc.) AND a documented history of inadequate response or intolerance to TCS and/or TCI.

Exclusion Criteria:

* Current or past history of other active skin diseases (e.g., psoriasis or Netherton syndrome or lupus erythematosus) or skin infections (bacterial, fungal, or viral) requiring systemic treatment within 4 weeks of the Baseline Visit or which would interfere with the appropriate assessment of AD lesions.
* Have used topical treatments for AD (except for topical emollient treatments) including but not limited to TCS, TCI, or topical phosphodiesterase type 4 (PDE-4) inhibitors, within 7 days of the Baseline Visit or any the following prohibited concomitant AD treatments within the specified timeframes below prior to the Baseline Visit:

  * Systemic therapy for AD, including but not limited to corticosteroids, methotrexate, cyclosporine, azathioprine, PDE-4 inhibitors, interferon-γ, and mycophenolate mofetil within 4 weeks;
  * Dupilumab within 8 weeks;
  * Targeted biologic treatments (other than dupilumab) within 5 half-lives (if known) or within 12 weeks, whichever is longer;
  * Phototherapy treatment, laser therapy, tanning booth, or extended sun exposure that could affect disease severity or interfere with disease assessments within 4 weeks.
* Known history of retinal detachment, previous cataract surgery, previous significant ocular trauma, or a known congenital ocular abnormality.
* For Randomized Cohort: diagnosed active parasitic infection; suspected or high risk of parasitic infection, unless clinical and (if necessary) laboratory assessment have ruled out active infection before randomization.

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 675 (Estimated)
Dates: Start 2024-08-19 (Actual); Primary Completion 2030-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving a 75% Reduction from Baseline in Eczema Area and Severity Index 75 (EASI 75) Score (other than US) | At Week 16
  EASI is a tool used to measure the extent (area) and severity of atopic eczema based on assessments of the head/neck, trunk, upper limbs and lower limbs. For each region the area score is recorded as the percentage of skin affected by eczema. For each region, the severity score is calculated as the sum of the intensity scores (scored as none [0], mild [1], moderate [2], or severe [3]) for redness (erythema, inflammation), thickness (induration, papulation, swelling - acute eczema), scratching (excoriation), and lichenification (lined skin, prurigo nodules - chronic eczema).
  The total EASI score for each region is calculated by multiplying the severity score by the area score, with adjustment for the proportion of the body region to the whole body. The final EASI score is the sum of the 4 region scores and ranges from 0 to 72 where higher scores represent worse disease.
Percentage of participants achieving validated Investigator Global Assessment for Atopic Dermatitis (vIGA-AD) 0 or 1 with a reduction from Baseline of ≥ 2 points (US and China only, descriptive) | Week 16
  The vIGA-AD is a validated assessment instrument to rate the severity of atopic dermatitis globally, based on the following scale:
  * 0 - Clear: No inflammatory signs of AD;
  * 1 - Almost clear: Barely perceptible erythema, induration/papulation and/or lichenification;
  * 2 - Mild: Slight but definite erythema, induration/papulation and/or minimal lichenification. No oozing or crusting;
  * 3 - Moderate: Clearly perceptible erythema, induration/papulation and/or lichenification, oozing or crusting may be present;
  * 4 - Severe: Marked erythema, induration/papulation and/or lichenification; Oozing or crusting may be present.
Number of Participants with Adverse Events (AEs) | Up to Approximately Week 172
  An AE is defined as any untoward medical occurrence in a patient or clinical investigation in which a participant is administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.

SECONDARY OUTCOMES:
Percentage of Participants Achieving a 75% Reduction from Baseline in EASI 75 Score (US) | At Week 16
  EASI is a tool used to measure the extent (area) and severity of atopic eczema based on assessments of the head/neck, trunk, upper limbs and lower limbs. For each region the area score is recorded as the percentage of skin affected by eczema. For each region, the severity score is calculated as the sum of the intensity scores (scored as none [0], mild [1], moderate [2], or severe [3]) for redness (erythema, inflammation), thickness (induration, papulation, swelling - acute eczema), scratching (excoriation), and lichenification (lined skin, prurigo nodules - chronic eczema).
  The total EASI score for each region is calculated by multiplying the severity score by the area score, with adjustment for the proportion of the body region to the whole body. The final EASI score is the sum of the 4 region scores and ranges from 0 to 72 where higher scores represent worse disease.
Percentage of participants achieving vIGA-AD of 0 or 1 (on a 5-point scale) with a reduction from Baseline of ≥ 2 Points | At Week 16
  The vIGA-AD is a validated assessment instrument to rate the severity of atopic dermatitis globally, based on the following scale:
  * 0 - Clear: No inflammatory signs of AD;
  * 1 - Almost clear: Barely perceptible erythema, induration/papulation and/or lichenification;
  * 2 - Mild: Slight but definite erythema, induration/papulation and/or minimal lichenification. No oozing or crusting;
  * 3 - Moderate: Clearly perceptible erythema, induration/papulation and/or lichenification, oozing or crusting may be present;
  * 4 - Severe: Marked erythema, induration/papulation and/or lichenification; Oozing or crusting may be present.
Percentage of participants achieving a 50% reduction from Baseline in EASI 50 score | At Week 16
  EASI is a tool used to measure the extent (area) and severity of atopic eczema based on assessments of the head/neck, trunk, upper limbs and lower limbs. For each region the area score is recorded as the percentage of skin affected by eczema. For each region, the severity score is calculated as the sum of the intensity scores (scored as none [0], mild [1], moderate [2], or severe [3]) for redness (erythema, inflammation), thickness (induration, papulation, swelling - acute eczema), scratching (excoriation), and lichenification (lined skin, prurigo nodules - chronic eczema).
  The total EASI score for each region is calculated by multiplying the severity score by the area score, with adjustment for the proportion of the body region to the whole body. The final EASI score is the sum of the 4 region scores and ranges from 0 to 72 where higher scores represent worse disease.
Percentage of participants achieving vIGA-AD of 0 or 1 (on a 5-point scale) with a reduction from Baseline of ≥ 2 Points | At Week 52
  The vIGA-AD is a validated assessment instrument to rate the severity of atopic dermatitis globally, based on the following scale:
  * 0 - Clear: No inflammatory signs of AD;
  * 1 - Almost clear: Barely perceptible erythema, induration/papulation and/or lichenification;
  * 2 - Mild: Slight but definite erythema, induration/papulation and/or minimal lichenification. No oozing or crusting;
  * 3 - Moderate: Clearly perceptible erythema, induration/papulation and/or lichenification, oozing or crusting may be present;
  * 4 - Severe: Marked erythema, induration/papulation and/or lichenification; Oozing or crusting may be present.
Percentage of participants achieving vIGA-AD of 0 or 1 (on a 5-point scale) with a reduction from Baseline of ≥ 2 Points | At Week 160
  The vIGA-AD is a validated assessment instrument to rate the severity of atopic dermatitis globally, based on the following scale:
  * 0 - Clear: No inflammatory signs of AD;
  * 1 - Almost clear: Barely perceptible erythema, induration/papulation and/or lichenification;
  * 2 - Mild: Slight but definite erythema, induration/papulation and/or minimal lichenification. No oozing or crusting;
  * 3 - Moderate: Clearly perceptible erythema, induration/papulation and/or lichenification, oozing or crusting may be present;
  * 4 - Severe: Marked erythema, induration/papulation and/or lichenification; Oozing or crusting may be present.
Percentage of participants achieving an improved (reduced) Patient Oriented Eczema Measure (POEM) of ≥ 4 points from from participants with POEM ≥ 4 at Baseline | At Week 16
  The POEM is a 7-item, validated questionnaire used to assess disease symptoms in both children and adults. Participants respond to 7 questions, including dryness, itching, flaking, cracking, sleep loss, bleeding, and weeping, each scored on a 5-point scale based on frequency of occurrence during the previous week: 0 = no days, 1 = 1 to 2 days, 2 = 3 to 4 days, 3 = 5 to 6 days, and 4 = all days. Item scores are added to provide a total score ranging from 0 (clear) to 28 (very severe atopic eczema). A change in POEM score of 3.4 points is considered the minimal clinically important difference.
Percentage of participants ≥ 4 years of age with a Baseline Children's Dermatology Life Quality Index (CDLQI) score of >1 achieving a CDLQI score of 0 or 1 | At Week 8
  The CDLQI is a 10-item, validated questionnaire used in clinical practice and clinical trials to assess the impact of dermatological disease symptoms and treatment on quality of life. The CDLQI has been validated for use in Participants 4 to 16 years of age. It consists of 10 questions assessing impact of skin diseases on different aspects of quality of life over the prior week. The CDLQI items include symptoms and feelings, daily activities, leisure, school, relationships, sleep, and treatment. Each item is scored on a 4-point scale: 0 = not at all; 1 = only a little; 2 = quite a lot; and 3 = very much. Item scores (0 to 3) are added to provide a total score range of 0 to 30; higher scores indicate greater impairment of quality of life.
Percentage of participants ≥ 4 years of age with a Baseline CDLQI score of >1 achieving a CDLQI score of 0 or 1 | At Week 16
  The CDLQI is a 10-item, validated questionnaire used in clinical practice and clinical trials to assess the impact of dermatological disease symptoms and treatment on quality of life. The CDLQI has been validated for use in Participants 4 to 16 years of age. It consists of 10 questions assessing impact of skin diseases on different aspects of quality of life over the prior week. The CDLQI items include symptoms and feelings, daily activities, leisure, school, relationships, sleep, and treatment. Each item is scored on a 4-point scale: 0 = not at all; 1 = only a little; 2 = quite a lot; and 3 = very much. Item scores (0 to 3) are added to provide a total score range of 0 to 30; higher scores indicate greater impairment of quality of life.
Percent change in Scoring Atopic Dermatitis (SCORAD) from Baseline | At Week 16
  SCORAD is a clinical tool used to assess the extent and severity of eczema (SCORing Atopic Dermatitis). The extent is assessed using the rule of 9 to calculate the affected area (A) as a percentage of the whole body (0-100%). The intensity part of the SCORAD (B) consists of 6 items: erythema, oedema/papulation, excoriations, lichenification, oozing/crusts and dryness, each graded on a scale from 0 (none) to 3 (severe), for a total score of 0 to 18. Subjective items (C) include daily pruritus and sleeplessness, each scored on a visual analogue scale (VAS) from 0 to 10 (total score 0-20). SCORAD is calculated as A/5 + 7B/2 + C, and ranges from 0 to 103 (worst). A negative change from Baseline indicates improvement.
Use of topical or systemic rescue therapy from Baseline to Week 16 | Baseline to Week 16
Number of days on rescue topical corticosteroid or topical calcineurin inhibitor from Baseline to Week 16 | Baseline to Week 16
Percentage of participants achieving a EASI 75 response for low dose upadacitinib daily adult equivalent dose | At Week 16
  EASI is a tool used to measure the extent (area) and severity of atopic eczema based on assessments of the head/neck, trunk, upper limbs and lower limbs. For each region the area score is recorded as the percentage of skin affected by eczema. For each region, the severity score is calculated as the sum of the intensity scores (scored as none [0], mild [1],
  An EASI 75 response is defined as a 75% reduction (improvement) from Baseline in EASI score.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (145):
- United States (29):
  - Applied Research Center Of Arkansas /ID# 268547, Little Rock, Arkansas
  - Integrative Skin Science and Research /ID# 265108, Sacramento, California
  - Clearlyderm Dermatology - West Boca /ID# 266323, Boca Raton, Florida
  - Pediatric Skin Research /ID# 266308, Coral Gables, Florida
  - Neoclinical Research - Hialeah /ID# 269694, Hialeah, Florida
  - Cleaver Medical Group Dermatology /ID# 265099, Dawsonville, Georgia
  - Aeroallergy Research Laboratory /ID# 267247, Savannah, Georgia
  - Treasure Valley Medical Research /ID# 266838, Boise, Idaho
  - Northwestern University Feinberg School of Medicine /ID# 265117, Chicago, Illinois
  - Sneeze Wheeze & Itch Associates /ID# 267238, Normal, Illinois
  - Dawes Fretzin, LLC /ID# 265097, Indianapolis, Indiana
  - Equity Medical, LLC /ID# 268270, Bowling Green, Kentucky
  - Maryland Allergy & Asthma Center /ID# 268032, Lanham, Maryland
  - DermAssociates - Rockville /ID# 266457, Rockville, Maryland
  - Washington University School of Medicine - St. Louis /ID# 268545, St Louis, Missouri
  - Skin Specialists /ID# 266331, Omaha, Nebraska
  - DOCS Clinical Research - Canal Winchester /ID# 268271, Canal Winchester, Ohio
  - Wright State Physicians Health Center /ID# 268841, Fairborn, Ohio
  - Oregon Health and Science University /ID# 266483, Portland, Oregon
  - Medical University of South Carolina /ID# 265113, Charleston, South Carolina
  - International Clinical Research - Tennessee /ID# 268548, Murfreesboro, Tennessee
  - Arlington Research Center, Inc /ID# 266330, Arlington, Texas
  - 3A Research - East location /ID# 267622, El Paso, Texas
  - Prime Clinical Research - Mansfield - East Broad Street /ID# 268042, Mansfield, Texas
  - Texas Dermatology and Laser Specialists /ID# 267249, San Antonio, Texas
  - Progressive Clinical Research - San Antonio /ID# 267262, San Antonio, Texas
  - Jordan Valley Dermatology & Research Center /ID# 267092, South Jordan, Utah
  - West Virginia University Hospitals /ID# 265114, Morgantown, West Virginia
  - Wisconsin Medical Center /ID# 267236, Milwaukee, Wisconsin
- Argentina (4):
  - Sanatorio 9 de Julio /ID# 267678, San Miguel de Tucumán, Tucumán Province
  - Conexa Investigacion Clinica /ID# 268728, Buenos Aires
  - Instituto de Neumonología y Dermatología /ID# 266146, Buenos Aires
  - Psoriahue - Buenos Aires /ID# 267737, Buenos Aires
- Australia (3):
  - The Children's Hospital at Westmead /ID# 265430, Westmead, New South Wales
  - Monash Health - Monash Medical Centre /ID# 267149, Clayton, Victoria
  - Institute for Skin, Health and Immunity /ID# 266158, Mitcham, Victoria
- Austria (3):
  - Medizinische Universitaet Graz /ID# 262741, Graz, Styria
  - Landeskrankenhaus Salzburg-Universitaetsklinikum der PMU (LKH) /ID# 265427, Salzburg
  - Medizinische Universitaet Wien /ID# 265417, Vienna
- Brazil (5):
  - Irmandade da Santa Casa de Misericórdia de Porto Alegre /ID# 267455, Porto Alegre, Rio Grande do Sul
  - Hospital e Maternidade Celso Pierro - PUC-Campinas /ID# 266965, Campinas, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina de Ribeirao Preto /ID# 266964, Ribeirão Preto, São Paulo
  - Clinica de Alergia Martti Antila /ID# 266197, Sorocaba, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao /ID# 266667, São Paulo
- Bulgaria (2):
  - UMHAT Alexandrovska EAD /ID# 265256, Sofiya, Sofia
  - Medical Center Cordis /ID# 265250, Pleven
- Canada (10):
  - Dermatology Research Institute - Blackfoot Trail /ID# 266744, Calgary, Alberta
  - Rejuvenation Dermatology - Edmonton Downtown /ID# 267871, Edmonton, Alberta
  - British Columbia Children and Women's Hospital and Health Centre /ID# 265395, Vancouver, British Columbia
  - Maritime Dermatology /ID# 267359, Halifax, Nova Scotia
  - Leader Research /ID# 266745, Hamilton, Ontario
  - Triple A Lab Inc /ID# 266615, Hamilton, Ontario
  - Lynderm Research Inc /ID# 267006, Markham, Ontario
  - Allergy Research Canada /ID# 270230, Niagara Falls, Ontario
  - DermAtelier on Avenue /ID# 267850, Toronto, Ontario
  - Centre Hospitalier Universitaire (CHU) Sainte-Justine /ID# 266831, Montreal, Quebec
- China (10):
  - Beijing Children's Hospital /ID# 266350, Beijing, Beijing Municipality
  - Children's Hospital Affiliated to Chongqing Medical University /ID# 266876, Yuzhong District, Chongqing Municipality
  - Xiamen Children's Hospital /ID# 266384, Xiamen, Fujian
  - Shenzhen Children's Hospital /ID# 266401, Shenzhen, Guangdong
  - Henan Children's Hospital Zhengzhou Children's Hospital /ID# 266832, Zhengzhou, Henan
  - Hunan Children's Hospital /ID# 266365, Changsha, Hunan
  - Dalian Women and Children's Medical Group /ID# 266675, Dalian, Liaoning
  - Chengdu Women and Children Center Hospital /ID# 266402, Chengdu, Sichuan
  - Kunming Childrens Hospital /ID# 266555, Kunming, Yunnan
  - The 2nd Affiliated Hospital and Yuying Children's Hospital of WMU /ID# 266708, Wenzhou, Zhejiang
- Croatia (5):
  - Klinika za dječje bolesti Zagreb /ID# 264936, Zagreb, City of Zagreb
  - Poliklinika DermaPlus /ID# 265724, Zagreb, City of Zagreb
  - Poliklinika Solmed /ID# 265070, Zagreb, City of Zagreb
  - Specialty Hospital Medico /ID# 266116, Rijeka, Primorje-Gorski Kotar County
  - Klinicki Bolnicki Centar KBC Split /ID# 265359, Split, Split-Dalmatia County
- France (8):
  - CHU Toulouse - Hopital Larrey /ID# 255048, Toulouse, Haute-Garonne
  - Centre Hospitalier Régional Universitaire de Nancy - Hôpitaux de Brabois /ID# 265455, Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - CHU Bordeaux - Hopital Pellegrin /ID# 266818, Bordeaux, Nouvelle-Aquitaine
  - Centre Hospitalier Universitaire de Nantes - L' Hopital l'hôtel-Dieu /ID# 265449, Nantes, Pays de la Loire Region
  - Centre Hospitalier Universitaire de Clermont Ferrand - Hopital Estaing /ID# 267327, Clermont-Ferrand, Puy-de-Dome
  - CHU Amiens-Picardie Site Sud /ID# 255083, Amiens, Somme
  - AP-HP - Hopital Necker /ID# 255050, Paris
  - Centre Hospitalier d Argenteuil Victor Dupouy /ID# 265448, Argenteuil, Île-de-France Region
- Germany (5):
  - Universitaetsklinikum Erlangen /ID# 255168, Erlangen, Bavaria
  - Fachklinik Bad Bentheim /ID# 255165, Bad Bentheim, Lower Saxony
  - Universitaetsklinikum Muenster /ID# 255166, Münster, North Rhine-Westphalia
  - Universitaetsklinikum Carl Gustav Carus Dresden /ID# 255167, Dresden, Saxony
  - Charite Universitaetsmedizin Berlin - Campus Mitte /ID# 267411, Berlin
- Hungary (3):
  - DermaMed Research - Oroshaza /ID# 266995, Orosháza, Bekes County
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont /ID# 265653, Szeged, Csongrád megye
  - Debreceni Egyetem-Klinikai Kozpont /ID# 265331, Debrecen, Hajdú-Bihar
- Israel (5):
  - Schneider Childrens Medical Center of Israel /ID# 265617, Petah Tikva, Central District
  - HaEmek Medical Center /ID# 266416, Afula, Haifa District
  - Hadassah Medical Center-Hebrew University /ID# 255041, Jerusalem, Jerusalem
  - Soroka Medical Center /ID# 265251, Beersheba, Southern District
  - The Chaim Sheba Medical Center /ID# 265254, Ramat Gan, Tel Aviv
- Italy (3):
  - Azienda Ospedaliero-Universitaria Policlinico Umberto I /ID# 267070, Rome, Roma
  - Ospedale Pediatrico Bambino Gesù /ID# 266118, Rome, Roma
  - IRCCS AOU di Bologna Policlinico Sant Orsola Malpighi /ID# 255118, Bologna
- Mexico (2):
  - Eukarya PharmaSite /ID# 265274, Monterrey, Nuevo León
  - Arke Smo Sa de Cv /Id# 266650, Veracruz
- Netherlands (2):
  - Amsterdam UMC, locatie AMC /ID# 265406, Amsterdam, North Holland
  - Erasmus Medisch Centrum /ID# 265408, Rotterdam, South Holland
- Poland (10):
  - Specjalistyczny Niepubliczny Zaklad Opieki Zdrowotnej Alergologia Plus /ID# 265457, Poznan, Greater Poland Voivodeship
  - MICS Centrum Medyczne Torun / Nasz Lekarz Przychodnie Medyczne /ID# 265454, Torun, Kuyavian-Pomeranian Voivodeship
  - Centrum Nowoczesnych Terapii Dobry Lekarz sp.z.o.o. /ID# 266030, Krakow, Lesser Poland Voivodeship
  - Klinika Osipowicz & Turkowski sp.z.o.o /ID# 267490, Warsaw, Masovian Voivodeship
  - Clinical Research Group Sp. z o.o. /ID# 266924, Warsaw, Masovian Voivodeship
  - Klinika Ambroziak Dermatologia /ID# 265458, Warsaw, Masovian Voivodeship
  - Royalderm Agnieszka Nawrocka /ID# 266606, Warsaw, Masovian Voivodeship
  - NZOZ Specjalistyczny Osrodek Dermatologiczny Dermal /ID# 266613, Bialystok, Podlaskie Voivodeship
  - Centrum Badan Klinicznych PI-House sp. z o.o. /ID# 265451, Gdansk, Pomeranian Voivodeship
  - Centrum Medyczne Angelius Provita /ID# 265456, Katowice, Silesian Voivodeship
- Portugal (3):
  - Unidade Local de Saude de Coimbra, EPE /ID# 266115, Coimbra
  - Unidade Local de Saude de Santo Antonio, E.P.E. /ID# 266112, Porto
  - Unidade Local de Saude Sao Joao, EPE /ID# 266111, Porto
- Puerto Rico (2):
  - Clinical Research Investigator Group, LLC /ID# 268366, Bayamón
  - Private Practice - Dr. Alma Cruz /ID# 264234, Carolina
- Singapore (2):
  - National University Hospital /ID# 265685, Singapore
  - KK Women's and Children's Hospital /ID# 266519, Singapore
- Slovakia (5):
  - Narodny Ustav Detskych Chorob /ID# 265253, Bratislava, Bratislava Region
  - ALERSA, s.r.o. /ID# 266245, Košice, Košice Region
  - Univerzitna nemocnica L. Pasteura Kosice /ID# 265239, Košice, Košice Region
  - Fakultna nemocnica Trnava /ID# 265245, Trnava
  - Univerzitna nemocnica Martin /ID# 265947, Martin, Žilina Region
- South Korea (6):
  - Korea University Ansan Hospital /ID# 264169, Ansan-si, Gyeonggido
  - Soon Chun Hyang University Hospital Bucheon /ID# 264171, Bucheon-si, Gyeonggido
  - Chungang University Hospital /ID# 266383, Dongjak-gu, Seoul Teugbyeolsi
  - Seoul National University Hospital /ID# 264176, Seoul, Seoul Teugbyeolsi
  - Konkuk University Medical Center /ID# 264178, Seoul, Seoul Teugbyeolsi
  - Hallym University Kangnam Sacred Heart Hospital /ID# 267318, Seoul, Seoul Teugbyeolsi
- Spain (5):
  - Hospital Sant Joan de Deu /ID# 255287, Esplugues de Llobregat, Barcelona
  - Hospital General Universitario Gregorio Maranon /ID# 255288, Madrid
  - Hospital Universitario La Paz /ID# 255286, Madrid
  - Consorci Hospital General Universitario de Valencia /ID# 255289, Valencia
  - Hospital Universitario Miguel Servet /ID# 255290, Zaragoza
- Taiwan (5):
  - Kaohsiung Chang Gung Memorial Hospital /ID# 267791, Kaohsiung City, Kaohsiung
  - New Taipei Municipal TuCheng Hospital (Built and Operated by Chang Gung Medical /ID# 266349, New Taipei City
  - National Taiwan University Hospital /ID# 265510, Taipei
  - Taipei Veterans General Hospital /ID# 265507, Taipei
  - Linkou Chang Gung Memorial Hospital /ID# 263664, Taoyuan
- United Kingdom (8):
  - Derriford Hospital and the Royal Eye Infirmary /ID# 266980, Plymouth, Devon
  - St Thomas' Hospital - Guy's and St Thomas' NHS Foundation Trust /ID# 265237, London, Greater London
  - Chelsea and Westminster Hospital /ID# 266389, London, Greater London
  - St George University Hospitals NHS Foundation Trust /ID# 266984, London, Greater London
  - University Hospital Southampton /ID# 266655, Southampton, Hampshire
  - Queen Elizabeth University Hospital - NHS Greater Glasgow and Clyde /ID# 265219, Glasgow, Lanarkshire
  - Manchester University NHS Foundation Trust /ID# 267693, Manchester
  - Royal Victoria Infirmary /ID# 265238, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M17-380